CLINICAL TRIAL: NCT01316328
Title: Determination of Predictive Genetic Markers of Toxicity After Hypofractionated Radiotherapy in Breast Cancer Patients Post-Conservative Surgery
Acronym: HYPOPRONE
Status: Completed | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Other Study IDs: IFO-84/10
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2010-12

CONDITIONS: Breast Cancer
Keywords: toxicity after single shot partial breast irradiation (SSPBI)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- BC patients after SSPBI: breast cancer (BC) patients following single shot partial breast irradiation (SSPBI) after breast conservative surgery

SUMMARY:
The single shot partial breast irradiation (SSPBI) trial was designed as a prospective Phase II "single-arm study". The use of a single dose tumor bed is expected to be very effective in terms of tumor control, but it could increase the incidence of radiation induced erythema. Therefore, the investigators assumed that a decreased DNA repair capability, as well as a reduced detoxification of the damage caused by oxidative stress could explain the increased acute toxicity, i.e. a higher incidence of erythema after a single dose. For this reason the investigators decided to investigate SNPs of genes involved in antioxidant and DNA damage repair pathways such as GST, XRCC1, XRCC3 and RAD51.

The investigators assumed an erythema rate of 20% and 54% in patient groups at low and high risk, respectively, (groups were identified based on the absence/presence of the above polymorphisms alone or in combination), thus the minimum sample size was 56 patients with α=0.05, 2-tailed test and a power of the study of 80%.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 48 years old with a life expectancy of at least 5 years
* Post-menopausal status
* Histologically proven, non lobular, adenocarcinoma of the breast

  * Primary tumours ≤ 3 cm
  * Negative surgical margins (≥ 2 mm)
  * Negative sentinel nodes or < 4 positive axillary nodes
  * No extra-capsular extension
* No previous radiotherapy

Exclusion Criteria:

* multicentric disease
* extended intraductal component (EIC > 25%)
* Paget's disease
* lobular adenocarcinoma
* distant metastases All the above criteria allow to identify patients at low risk of local recurrence.

Ages: 48 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer (BC) patients following single shot partial breast irradiation(SSPBI) after breast conservative surgery
Sampling Method: Non-Probability Sample
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Elena NCI, Rome, Rome, Italy

REFERENCES:
- [Derived] Falvo E, Strigari L, Citro G, Giordano C, Boboc G, Fabretti F, Bruzzaniti V, Bellesi L, Muti P, Blandino G, Pinnaro P. SNPs in DNA repair or oxidative stress genes and late subcutaneous fibrosis in patients following single shot partial breast irradiation. J Exp Clin Cancer Res. 2012 Jan 24;31(1):7. doi: 10.1186/1756-9966-31-7. PMID 22272830
- [Derived] Pinnaro P, Arcangeli S, Giordano C, Arcangeli G, Impiombato FA, Pinzi V, Iaccarino G, Soriani A, Landoni V, Strigari L. Toxicity and cosmesis outcomes after single fraction partial breast irradiation in early stage breast cancer. Radiat Oncol. 2011 Nov 11;6:155. doi: 10.1186/1748-717X-6-155. PMID 22079051
- [Derived] Falvo E, Strigari L, Citro G, Giordano C, Arcangeli S, Soriani A, D'Alessio D, Muti P, Blandino G, Sperduti I, Pinnaro P. Dose and polymorphic genes xrcc1, xrcc3, gst play a role in the risk of articledeveloping erythema in breast cancer patients following single shot partial breast irradiation after conservative surgery. BMC Cancer. 2011 Jul 12;11:291. doi: 10.1186/1471-2407-11-291. PMID 21749698